CLINICAL TRIAL: NCT02172560
Title: A Retrospective Collection of Vital Status and Pulmonary Medication Usage Data for Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Withdrew Prematurely From Either of Two One-Year Trials (205.254, 205.255) of Tiotropium Inhalation Solution Delivered by the Respimat Inhaler
Brief Title: A Collection of Vital Status and Pulmonary Medication Usage Data for Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Withdrew Prematurely From Tiotropium Inhalation Solution Delivered by the Respimat Inhaler
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.392
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Premature withdrawal from tiotropium
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium

SUMMARY:
The objectives were to collect information on vital status and pulmonary medication use at the predicted exit date for patients who participated in two one-year trials and withdrew prematurely. The primary objective was to ascertain the vital status (dead or alive) of these patients in the time interval between the patients' withdrawal from the trial and their predicted exit date (i.e: 48 weeks from first intake of randomised treatment + 30 days). The secondary objective was to collect information on classes of pulmonary medication and some other specified pulmonary interventions used by these prematurely discontinued patients at the time of their predicted exit date (i.e 48 weeks from the first intake of randomised treatment + 30 days) or at date of death (if this occurred during the time interval of interest, i.e 48 weeks from the first intake of randomised treatment + 30 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients who withdrew prematurely from the randomised treatment phase of studies 205.254 and 205.255.

Exclusion Criteria:

* Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COPD who withdrew prematurely from the randomised treatment phases of studies 205.254 and 205.255
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number and status of patients dead or alive at the predicted end of treatment date | Until 48 weeks after first intake of randomised treatment + 30 days follow-up or date of death

SECONDARY OUTCOMES:
Number and specification of patients on pulmonary medications and other pulmonary interventions | Until 48 weeks after first intake of randomised treatment + 30 days follow-up or date of death

CONTACTS AND LOCATIONS:
Locations (19):
- Australia (7):
  - Boehringer Ingelheim Investigational Site 61501, Garran, Australian Capital Territory
  - Boehringer Ingelheim Investigational Site 61403, Clayton, New South Wales
  - Boehringer Ingelheim Investigational Site 61502, Adelaide, South Australia
  - Boehringer Ingelheim Investigational Site 61401, Woodsville South, South Australia
  - Boehringer Ingelheim Investigational Site 61402, Frankston, Victoria
  - Boehringer Ingelheim Investigational Site 61503, Nedlands, Western Australia
  - Boehringer Ingelheim Investigational Site 61405, Perth, Western Australia
- New Zealand (2):
  - Boehringer Ingelheim Investigational Site 61505, Hamilton
  - Boehringer Ingelheim Investigational Site 61504, Otahuhu
- United Kingdom (10):
  - Boehringer Ingelheim Investigational Site 44402, Birmingham
  - Boehringer Ingelheim Investigational Site 44409, Bristol
  - Boehringer Ingelheim Investigational Site 44502, Devon
  - Boehringer Ingelheim Investigational Site 44504, Hull
  - Boehringer Ingelheim Investigational Site 44507, Isleworth
  - Boehringer Ingelheim Investigational Site 44506, Manchester
  - Boehringer Ingelheim Investigational Site 44403, Nottingham
  - Boehringer Ingelheim Investigational Site 44405, Swansea
  - Boehringer Ingelheim Investigational Site 44404, Torquay
  - Boehringer Ingelheim Investigational Site 44505, Torquay